CLINICAL TRIAL: NCT03337425
Title: Psychoeducational Groups for Adults With Attention-Deficit Hyperactivity/Impulsivity Disorder (ADHD): a Randomized Waitlist-controlled Multicenter Pilot Trial
Brief Title: Psychoeducational Groups for Adults With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1885
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Psychotherapy, group; Adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Waiting Lists; Therapeutics

STUDY DESIGN:
Intervention Model Description: a Norwegian multicenter study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psychoeducational groups (Experimental): Psychoeducational group therapy and standard treatment (ADHD treatment as usual)
  Interventions: Behavioral: Psychoeducational group therapy; Other: Standard treatment
- Waiting list (Active Comparator): Waiting list and standard treatment (ADHD treatment as usual)
  Interventions: Behavioral: Waiting list; Other: Standard treatment

INTERVENTIONS:
Behavioral: Psychoeducational group therapy — The group-based psychoeducational program consists of 10 sessions, run over 10 consecutive weeks. Each session consist of a lecture, given by a recruited expert on the topic of the session (20 minutes) with a following discussion of the topic (45 minutes), facilitated by the course leader. All sessions are organized and led by the course leader, which also includes keeping structure in time, discussion and closing of the session. Psychoeducation comes in addition to standard treatment (ADHD treatment as usual).
  Arms: psychoeducational groups
Behavioral: Waiting list — Waiting list and standard treatment (ADHD treatment as usual)
  Arms: Waiting list
Other: Standard treatment — Standard treatment consists of diagnostic assessment of ADHD and comorbidity, as well as treatment with medication. In addition, some patients receive cognitive behavioral therapy, although this is not systematically given to every patient. If needed, patients are also offered assistance with regard to economy, housing, education and work. As well as contact with family and network.
  Other Names: Treatment as usual

SUMMARY:
This pilot study aims to assess patient satisfaction and preliminary efficacy of a psychoeducational group treatment, using a randomized waitlist-controlled trial, at two different outpatient clinics in mid-Norway. All participants will receive standard treatment during the intervention period. Assessment of client satisfaction (CSQ 8), general self-efficacy (GSE-6), ADHD-related quality of life (AAQoL) symptoms of ADHD (SCL-9; ASRS), and work participation will be conducted at time of recruitment prior to randomization (T0), pre- (T1), post-treatment (T2), with a 10 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* confirmed ADHD diagnosis
* speaking a Scandinavian language

Exclusion Criteria:

* not able or willing to give informed consent
* psychosis
* severe learning difficulties

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change in patient satisfaction | Baseline, post-intervention (10 weeks) and after 10 weeks follow-up (20 weeks)
  Measured with a modified version of the Client Satisfaction Questionnaire (CSQ-8). The scale consists of 8 items measured on a scale from 1 to 4. A sum score between 8 and 32 indicate the level of satisfaction with services provided.
Change in general self-efficacy | Baseline, post-intervention (10 weeks) and after 10 weeks follow-up (20 weeks)
  Measured with General Self-Efficacy Scale (GSE-6), a short-form measure of self-efficacy. Self-efficacy is regarded as a protective factor in adapting to stress and chronic illness. The scale consists of 6 items, measured on a 4-point scale, with a possible range of 6-24.

SECONDARY OUTCOMES:
Change in ADHD-related symptoms (ASRS) | Baseline, post-intervention (10 weeks) and after 10 weeks follow-up (20 weeks)
  Measured with ASRS, a self-reporting scale for ADHD-related symptoms in adults. The scale consists of 18 items, based on DSM-V diagnostic criteria for ADHD. The items are measured on a 5-point scale, with a possible range of 0-72.
Change in ADHD-related symptoms (SCL-9) | Baseline, post-intervention (10 weeks) and after 10 weeks follow-up (20 weeks)
  Measured with 9 items from the SCL-90. SCL-9 is an ADHD-specific scale, consisting of 9 items of the original 90. SCL-9 covers the specific characteristic traits of ADHD.
Change in ADHD-related quality of life | Baseline, post-intervention (10 weeks) and after 10 weeks follow-up (20 weeks)
  Measured with AAQoL - which covers ADHD-specific quality of life and function. AAQoL consists of 29 questions measuring health related quality of life among adults with ADHD.

CONTACTS AND LOCATIONS:
Overall Officials: Terje Torgersen, phd, Principal Investigator — St. Olavs Hospital
Locations (2):
- Norway (2):
  - Levanger Hospital, Nord-Trøndelag Hospital Trust, Levanger, N-T
  - Tiller DPS - St. Olavs University Hospital, Trondheim, S-T

REFERENCES:
- [Background] Vaag JR, Lara-Cabrera ML, Hjemdal O, Gjervan B, Torgersen T. Psychoeducational groups versus waitlist in treatment of attention-deficit hyperactivity/impulsivity disorder (ADHD) in adults: a protocol for a pilot randomized waitlist-controlled multicenter trial. Pilot Feasibility Stud. 2019 Jan 23;5:17. doi: 10.1186/s40814-019-0401-1. eCollection 2019. PMID 30693097
- [Derived] Holsbrekken A, Skliarova T, Mandahl A, Saether SG, Lund AGS, Surkovic J, Sondenaa E, Vaag J, Torgersen T, Lara-Cabrera ML. Effects of a psychoeducational group intervention for adults diagnosed with ADHD: a pilot randomized controlled study. BMC Psychiatry. 2025 Oct 14;25(1):983. doi: 10.1186/s12888-025-07452-5. PMID 41088068